CLINICAL TRIAL: NCT00485056
Title: Pioglitazone on Cardiac Function and Large Arteries (PICCOLA)
Brief Title: Pioglitazone on Cardiac Function and Large Arteries (PICCOLA Study)
Acronym: PICCOLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EU-IIT-006
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes
Keywords: Diabetes; Tissue doppler imaging; Wave intensity analysis.
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Crossover arm
  Interventions: Drug: Pioglitazone
- Pioglitazone (Active Comparator): Pioglitazone 45mgs daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 45mgs daily

SUMMARY:
This study aims to use a novel, sensitive, non-invasive scanning technique to investigate the effects of insulin-sensitizing agent pioglitazone, on heart and artery function.

DETAILED DESCRIPTION:
The prevalence of diabetes mellitus and impaired glucose tolerance are nearing epidemic proportions in developed societies. For example in the USA >16 million individuals have diabetes and this number is predicted to double over the next two decades. Diabetes is a major risk factor for death and disability, primarily from cardiovascular disease (CVD).

The mechanisms of how diabetes increases the risk of developing CVD are not fully understood. It is evident from previous studies that diabetes has an adverse effect on both artery and heart function. What is emerging from recent studies is that it is likely that these proven dysfunctions in the arteries and heart interact to increase the risk of CVD.

Insulin-sensitizing agents, such as Pioglitazone, may have a beneficial effect on heart and artery function. This study aims to further our understanding of the effect of these agents on heart and artery using a novel, sensitive, non-invasive scanning technique to investigate the effects of this group of drugs on heart and artery function.

This is a prospective double-blind randomised crossover study comparing the insulin-sensitizing drug, Pioglitazone with a placebo in 24 volunteers. Following a >1 week run-in period subjects will be randomised double-blind to 1 of 2 treatment sequences. Subjects will either receive the active drug (Pioglitazone 45mg/day) for a 12 week period, followed by a 2 week washout and then the placebo drug for 12 weeks OR they will receive the placebo drug for 12 weeks, followed by the 2 week washout and 12 weeks of the active drug (Pioglitazone 45mg/day).

This design was chosen to test the null hypothesis that the active drug will have no effect on diastolic heart function. The use of a placebo is essential to ensure that any benefits found can be attributed to the active drug. The design also allows us to minimise the number of subjects needed and is the gold standard approach to avoid observer bias.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age with Type 2 Diabetes

Exclusion Criteria:

* Subjects will be excluded if they have any of the following:

  * Known coronary heart disease,
  * Patients receiving Insulin,
  * Uncontrolled hypertension (i.e. >160mmHg systolic or >95mmHg diastolic),
  * Systolic dysfunction (ejection fraction <50%),
  * Heart Valve Disease,
  * Proliferative or pre-proliferative retinopathy,
  * Severe hepatic or renal impairment.
  * Possible pregnancy
  * Malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the TDI E' ratio which is the relatively preload independent measure of ventricular diastolic function. | 26 weeks

SECONDARY OUTCOMES:
E/E' measured by TDI (a non-invasive measure of preload). | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alun D Hughes, phd, Principal Investigator — Imperial College London
Locations (1):
- International Centre for Circulatory Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No